CLINICAL TRIAL: NCT02287909
Title: Pharmacodynamic Evaluation of Switching From Ticagrelor to Clopidogrel in Patients With Coronary Artery Disease
Brief Title: Switching From Ticagrelor to Clopidogrel in Patients With Coronary Artery Disease
Acronym: SWAP-4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFJ 2014-153
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- A) clopidogrel 600 mg LD 24 hours after last MD of ticagrelor (Experimental): Patients will be randomized (1:1:1:1) into one of the four following groups: A) clopidogrel 600 mg LD 24 hours after last MD of ticagrelor, followed by 75mg daily MD; B) clopidogrel 600 mg LD 12 hours after last MD of ticagrelor, followed by 75mg daily MD; C) clopidogrel 75mg daily MD 24 hours after last MD of ticagrelor; D) continue ticagrelor MD 90mg twice daily
  Interventions: Drug: Clopidogrel
- B) clopidogrel 600 mg LD 12 hours after last MD of ticagrelor (Experimental): Patients will be randomized (1:1:1:1) into one of the four following groups: A) clopidogrel 600 mg LD 24 hours after last MD of ticagrelor, followed by 75mg daily MD; B) clopidogrel 600 mg LD 12 hours after last MD of ticagrelor, followed by 75mg daily MD; C) clopidogrel 75mg daily MD 24 hours after last MD of ticagrelor; D) continue ticagrelor MD 90mg twice daily
  Interventions: Drug: Clopidogrel
- C) clopidogrel 75mg MD 24 hours after last MD of ticagrelor (Experimental): Patients will be randomized (1:1:1:1) into one of the four following groups: A) clopidogrel 600 mg LD 24 hours after last MD of ticagrelor, followed by 75mg daily MD; B) clopidogrel 600 mg LD 12 hours after last MD of ticagrelor, followed by 75mg daily MD; C) clopidogrel 75mg daily MD 24 hours after last MD of ticagrelor; D) continue ticagrelor MD 90mg twice daily
  Interventions: Drug: Clopidogrel
- D) continue ticagrelor MD 90mg twice daily (Active Comparator): Patients will be randomized (1:1:1:1) into one of the four following groups: A) clopidogrel 600 mg LD 24 hours after last MD of ticagrelor, followed by 75mg daily MD; B) clopidogrel 600 mg LD 12 hours after last MD of ticagrelor, followed by 75mg daily MD; C) clopidogrel 75mg daily MD 24 hours after last MD of ticagrelor; D) continue ticagrelor MD 90mg twice daily
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel — Swiching from ticagrelor to clopidogrel
  Other Names: Plavix
  Arms: A) clopidogrel 600 mg LD 24 hours after last MD of ticagrelor; B) clopidogrel 600 mg LD 12 hours after last MD of ticagrelor; C) clopidogrel 75mg MD 24 hours after last MD of ticagrelor
Drug: Ticagrelor — Continue treatment with ticagrelor
  Other Names: Brilinta
  Arms: D) continue ticagrelor MD 90mg twice daily

SUMMARY:
The recommended antiplatelet treatment regimen for patients affected by acute coronary syndromes (ACS) and those undergoing percutaneous coronary intervention (PCI) consists in the combination of aspirin and a P2Y12 receptor inhibitor. More potent P2Y12 receptor inhibitors, such as ticagrelor, have been developed which are associated with less response variability than clopidogrel and better clinical outcomes. Ticagrelor use has increased significantly because of its more expanded Food and Drug Administration (FDA) indications compared with prasugrel. However, despite the evidence for sustained efficacy and safety, many physicians limit treatment duration with ticagrelor to the early phases following an ACS mostly due to cost issues and concerns about increased bleeding. Therefore, it is very common in clinical practice to switch patients while on maintenance dosing (MD) with ticagrelor to treatment with clopidogrel. However, the pharmacodynamic (PD) effects of switching from ticagrelor to clopidogrel remain unknown. Therefore, the aim of this investigation is to evaluate the PD effects of switching from ticagrelor to clopidogrel.

DETAILED DESCRIPTION:
The recommended antiplatelet treatment regimen for patients affected by acute coronary syndromes (ACS) and those undergoing percutaneous coronary intervention (PCI) consists in the combination of aspirin and a P2Y12 receptor inhibitor. Currently, three P2Y12 receptor inhibitors are available for clinical use (clopidogrel, prasugrel, and ticagrelor). Among these, clopidogrel remains the most widely used. However, recent studies have shown that there is a broad variability in platelet-inhibitory response induced by clopidogrel, which in turn is associated with worse outcomes. More potent P2Y12 receptor inhibitors (prasugrel and ticagrelor) have been developed which are associated with less response variability than clopidogrel and better clinical outcomes. Ticagrelor use has increased significantly because of its more expanded Food and Drug Administration (FDA) indications compared with prasugrel. However, despite the evidence for sustained efficacy and safety, many physicians limit treatment duration with ticagrelor to the early phases following an ACS (early weeks or months, rather than one-year) mostly due to cost issues and concerns about increased bleeding. Therefore, it is very common in clinical practice to switch patients while on maintenance dosing (MD) with ticagrelor to treatment with clopidogrel. However, the pharmacodynamic (PD) effects of switching from ticagrelor to clopidogrel remain unknown. In addition, it is unknown whether switching from ticagrelor to clopidogrel should occur with or without a loading dose (LD). Therefore, the aim of this investigation is to evaluate the PD effects of switching from ticagrelor to clopidogrel with and without a LD. The present study has a prospective, randomized, open-label design, in which patients will be treated with 4 different strategies to assess PD profiling after switching. This study will provide important insights on PD effects of switching from ticagrelor to clopidogrel.

ELIGIBILITY:
Inclusion Criteria

1. Patients with angiographically documented CAD
2. On therapy with aspirin(<100mg/day) and clopidogrel (75mg/day) for at least 30 days per standard of care
3. Age between 18 and 80 years old

Exclusion Criteria

1. History of intracranial bleeding
2. Severe hepatic impairment (ALT >2.5 times the upper limit of normal)
3. Active bleeding or propensity to bleed or blood dycrasia
4. Platelet count <80x106/mL
5. Hemoglobin <10g/dL
6. Hemodynamic instability
7. Estimated glomerular filtration rate (eGFR) <30 mL/min
8. On treatment with oral anticoagulants
9. Patients with sick sinus syndrome (SSS) or II or III degree AV block without pacemaker protection
10. Drugs interfering CYP3A4 metabolism (to avoid interaction with ticagrelor): ketoconazole, itraconazole, voriconazole, clarithromicin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir and telithromizycin
11. Pregnant females [women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study].

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Angiolillo, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Franchi F, Rollini F, Rivas Rios J, Rivas A, Agarwal M, Kureti M, Nagaraju D, Wali M, Shaikh Z, Briceno M, Nawaz A, Moon JY, Been L, Suryadevara S, Soffer D, Zenni MM, Bass TA, Angiolillo DJ. Pharmacodynamic Effects of Switching From Ticagrelor to Clopidogrel in Patients With Coronary Artery Disease: Results of the SWAP-4 Study. Circulation. 2018 Jun 5;137(23):2450-2462. doi: 10.1161/CIRCULATIONAHA.118.033983. Epub 2018 Mar 11. PMID 29526833

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 87 patients entered a run-in phase. Of these, 7 withdrew during run in.
Period: Overall Study
Arm/Group | A) Clopidogrel 600 mg LD 24 Hours After Last MD of Ticagrelor | B) Clopidogrel 600 mg LD 12 Hours After Last MD of Ticagrelor | C) Clopidogrel 75mg MD 24 Hours After Last MD of Ticagrelor | D) Continue Ticagrelor MD 90mg Twice Daily
Started | 20 | 20 | 20 | 20
Completed | 18 | 19 | 20 | 19
Not Completed | 2 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A) Clopidogrel 600 mg LD 24 Hours After Last MD of Ticagrelor | B) Clopidogrel 600 mg LD 12 Hours After Last MD of Ticagrelor | C) Clopidogrel 75mg MD 24 Hours After Last MD of Ticagrelor | D) Continue Ticagrelor MD 90mg Twice Daily | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: information for each of the 4 groups and overall provided and mean and SD
  years | 62 (7) | 65 (8) | 63 (9) | 58 (9) | 62 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 7 | 8 | 29
  Male | 11 | 15 | 13 | 12 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 5 | 7 | 6 | 28
  White | 10 | 14 | 13 | 14 | 51
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 20 | 20

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity Unit
Description: PRU assessed by VerifyNow at 48 hours after switching of clopidogrel 600 mg LD administered 24 hours after the last ticagrelor MD vs. clopidogrel 75 mg MD given 24 hours after the last ticagrelor MD
Time Frame: 48 hours after switch
Measure: Least Squares Mean (Standard Error); unit: PRU
Arm/Group | A) Clopidogrel 600 mg LD 24 Hours After Last MD of Ticagrelor | B) Clopidogrel 600 mg LD 12 Hours After Last MD of Ticagrelor | C) Clopidogrel 75mg MD 24 Hours After Last MD of Ticagrelor | D) Continue Ticagrelor MD 90mg Twice Daily
Number analyzed (Participants) | 18 | 19 | 20 | 19
PRU | 177 (27) | 164 (24) | 174 (24) | 26 (25)
Statistical Analysis 1: Comparison: A) Clopidogrel 600 mg LD 24 Hours After Last MD of Ticagrelor vs C) Clopidogrel 75mg MD 24 Hours After Last MD of Ticagrelor; Test type: Superiority; p > 0.05, ANCOVA; least square mean difference = -6.9, 985% CI 2-sided [-38 to 24]

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | A) Clopidogrel 600 mg LD 24 Hours After Last MD of Ticagrelor | B) Clopidogrel 600 mg LD 12 Hours After Last MD of Ticagrelor | C) Clopidogrel 75mg MD 24 Hours After Last MD of Ticagrelor | D) Continue Ticagrelor MD 90mg Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 0/20 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A) Clopidogrel 600 mg LD 24 Hours After Last MD of Ticagrelor (N=20) | B) Clopidogrel 600 mg LD 12 Hours After Last MD of Ticagrelor (N=20) | C) Clopidogrel 75mg MD 24 Hours After Last MD of Ticagrelor (N=20) | D) Continue Ticagrelor MD 90mg Twice Daily (N=20)
Dypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Dyspnea
Bleeding (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — BARC 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT02287909/Prot_SAP_000.pdf